CLINICAL TRIAL: NCT02979626
Title: Evaluation of Moderate to Severe Influenza Disease in Children 6 Months to 8 Years in Colorado
Brief Title: Evaluation of Moderate to Severe Influenza Outcomes in Children
Acronym: M2SFlu
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-1785
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Influenza; Otitis Media; Lower Resp Tract Infection; Encephalitic Infection; Myositis Viral; Fever
Keywords: hospitalization; intensive care unit; school absenteeism; work absenteeism
MeSH Terms: conditions — Influenza, Human; Otitis Media; Encephalitis; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Respiratory swab samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Moderate-to-severe Influenza: Children 6 weeks to 8 years of age with influenza-like illness and one of the following:
  1. Fever >39
  2. Lower respiratory tract infection
  3. Acute otitis media
  4. Serious extra-pulmonary manifestations (myositis, encephalitis)
  Interventions: Procedure: Respiratory nasal swab
- Mild Influenza: Children 6 weeks to 8 years of age with influenza-like illness (ILI) without the criteria for moderate-to-severe disease (above)
  Interventions: Procedure: Respiratory nasal swab

INTERVENTIONS:
Procedure: Respiratory nasal swab — Nasal swabs will be obtained for testing by the study nurses. If a respiratory sample has already been collected as part of routine clinical care, this will replace the study collection, and no additional testing will be required.
  Other Names: Nasal swab

SUMMARY:
The purpose of this study was to determine whether moderate-severe endpoints (including high fever, lower respiratory tract disease, acute otitis media, or serious extra-pulmonary complications) were predictive of hospitalization, intensive care admission, antibiotic use and other complications in children under 8 years of age.

DETAILED DESCRIPTION:
This prospective observational study aimed to determine the risk difference of hospitalization due to moderate to severe influenza compared with mild influenza among children aged 6 months to 8 years who were evaluated at Children's Hospital Colorado emergency department and urgent care during the 2016-2017 influenza season. In addition, the study intended to evaluate the risk difference for other health outcomes such as ICU admission, antibiotic and antiviral use, caregiver and child absenteeism and recurrent (>1) healthcare visits, and to compare the healthcare costs associated with management of moderate to severe versus mild influenza in children. Children who presented to Children's Hospital Colorado Emergency Department (ED) and urgent care affiliated sites (North Campus urgent care) with an influenza-like illness from December 2016 to April 2017 and during the 2016-2017 influenza season, were eligible for the study. Once enrolled in the study, the investigators collected respiratory samples (nasal swab specimens) for influenza testing by PCR, sociodemographic and clinical data including variables of interest outlined above, and followed the clinical outcome of these children for 14 days after their initial presentation. Some of the variables of interest the investigators collected are shown below.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to < 8 years
* Presentation to one of the study sites with signs and symptoms of influenza-like illness (temperature of >37.8⁰C and at least one of the following: cough, sore throat, runny nose or nasal congestion)
* Parents or guardians agreeing and consenting to medical information release, respiratory specimen collection and testing, email/phone call follow up and collection of leftover blood samples obtained during routine clinical care
* Patients seen during the 2016-2017 influenza season

Exclusion Criteria:

* Respiratory symptom duration > 14 days
* Nurse only visit
* Enrollment in the study within prior 14 days

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 6 months to 8 years of age and younger seeking evaluation and management of influenza-like illness (ILI) at any of the study sites will be eligible for participation in the study. The study will commence during the influenza season as determined by the department of microbiology and epidemiology at CHCO (the influenza season commences when there are 3 positive influenza PCR tests within a week), approximately from December 1, 2016 to April 30, 2017.
Sampling Method: Non-Probability Sample
Enrollment: 1478 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin J Asturias, MD, Principal Investigator — University of Colorado, Denver; Suchitra Rao, MD, Study Director — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Hospital North Campus Urgent Care, Broomfield, Colorado

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilkes JJ, Leckerman KH, Coffin SE, Keren R, Metjian TA, Hodinka RL, Zaoutis TE. Use of antibiotics in children hospitalized with community-acquired, laboratory-confirmed influenza. J Pediatr. 2009 Mar;154(3):447-9. doi: 10.1016/j.jpeds.2008.09.026. PMID 19874761
- [Background] Coffin SE, Zaoutis TE, Rosenquist AB, Heydon K, Herrera G, Bridges CB, Watson B, Localio R, Hodinka RL, Keren R. Incidence, complications, and risk factors for prolonged stay in children hospitalized with community-acquired influenza. Pediatrics. 2007 Apr;119(4):740-8. doi: 10.1542/peds.2006-2679. PMID 17403845
- [Background] Izurieta HS, Thompson WW, Kramarz P, Shay DK, Davis RL, DeStefano F, Black S, Shinefield H, Fukuda K. Influenza and the rates of hospitalization for respiratory disease among infants and young children. N Engl J Med. 2000 Jan 27;342(4):232-9. doi: 10.1056/NEJM200001273420402. PMID 10648764
- [Background] Neuzil KM, Mellen BG, Wright PF, Mitchel EF Jr, Griffin MR. The effect of influenza on hospitalizations, outpatient visits, and courses of antibiotics in children. N Engl J Med. 2000 Jan 27;342(4):225-31. doi: 10.1056/NEJM200001273420401. PMID 10648763
- [Background] Salo H, Kilpi T, Sintonen H, Linna M, Peltola V, Heikkinen T. Cost-effectiveness of influenza vaccination of healthy children. Vaccine. 2006 Jun 5;24(23):4934-41. doi: 10.1016/j.vaccine.2006.03.057. Epub 2006 Apr 7. PMID 16678945
- [Background] Ferdinands JM, Olsho LE, Agan AA, Bhat N, Sullivan RM, Hall M, Mourani PM, Thompson M, Randolph AG; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Effectiveness of influenza vaccine against life-threatening RT-PCR-confirmed influenza illness in US children, 2010-2012. J Infect Dis. 2014 Sep 1;210(5):674-83. doi: 10.1093/infdis/jiu185. Epub 2014 Mar 26. PMID 24676207
- [Background] Heikkinen T, Silvennoinen H, Heinonen S, Vuorinen T. Clinical and socioeconomic impact of moderate-to-severe versus mild influenza in children. Eur J Clin Microbiol Infect Dis. 2016 Jul;35(7):1107-13. doi: 10.1007/s10096-016-2641-9. Epub 2016 Apr 16. PMID 27086364
- [Background] Jain VK, Rivera L, Zaman K, Espos RA Jr, Sirivichayakul C, Quiambao BP, Rivera-Medina DM, Kerdpanich P, Ceyhan M, Dinleyici EC, Cravioto A, Yunus M, Chanthavanich P, Limkittikul K, Kurugol Z, Alhan E, Caplanusi A, Durviaux S, Boutet P, Ofori-Anyinam O, Chandrasekaran V, Dbaibo G, Innis BL. Vaccine for prevention of mild and moderate-to-severe influenza in children. N Engl J Med. 2013 Dec 26;369(26):2481-91. doi: 10.1056/NEJMoa1215817. Epub 2013 Dec 11. PMID 24328444
- [Derived] Rao S, Moss A, Lamb M, Innis BL, Asturias EJ. Vital sign predictors of severe influenza among children in an emergent care setting. PLoS One. 2022 Aug 12;17(8):e0272029. doi: 10.1371/journal.pone.0272029. eCollection 2022. PMID 35960719
- [Derived] Rao S, Moss A, Lamb MM, Asturias EJ. Evaluation of Influenza Vaccine Effectiveness Among Young Children Receiving Consecutive Versus Nonconsecutive Vaccination During Influenza A(H3N2)-Predominant Seasons. J Pediatric Infect Dis Soc. 2021 Apr 3;10(3):359-362. doi: 10.1093/jpids/piaa080. PMID 32756876
- [Derived] Rao S, Yanni E, Moss A, Lamb MM, Schuind A, Bekkat-Berkani R, Innis BL, Cotter J, Mistry RD, Asturias EJ. Evaluation of a New Clinical Endpoint for Moderate to Severe Influenza Disease in Children: A Prospective Cohort Study. J Pediatric Infect Dis Soc. 2020 Sep 17;9(4):460-467. doi: 10.1093/jpids/piz075. PMID 31724050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from January 30, 2017 until 5 May of 2018 including 2 influenza seasons at the Children's Hospital Colorado main Emergency Department and a peripheral Urgent Care Center
Groups:
- Moderate-to-severe Influenza: Children 6 weeks to 8 years of age with influenza-like illness and one of the following:
  1. Fever >39
  2. Lower respiratory tract infection
  3. Acute otitis media
  4. Serious extra-pulmonary manifestations (myositis, encephalitis)
  Respiratory nasal swab: Nasal swabs will be obtained for testing by the study nurses. If a respiratory sample has already been collected as part of routine clinical care, this will replace the study collection, and no additional testing will be required.
Period: Overall Study
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Started | 313 | 98
Completed | 313 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Influenza positive ONLY
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate-to-severe Influenza | Mild Influenza | Total
Number analyzed (Participants) | 313 | 98 | 411
Age, Continuous [Median (Standard Deviation); unit: years] — Population: Subjects analyzed are ONLY influenza positive confirmed
  years | 3.8 (1.8) | 4.8 (2.4) | 4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 53 | 205
  Male | 161 | 45 | 206
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 14 | 38
  White | 93 | 15 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 196 | 69 | 265

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization
Description: Hospitalization within 14 days of influenza infection diagnosis
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 313 | 98
Participants | 26 | 2

2. Secondary Outcome: ICU Admission
Description: Admission to the intensive care unit after influenza diagnosis
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 313 | 98
Participants | 3 | 0

3. Secondary Outcome: Antiviral Use
Description: Antiviral use in children presenting to the ED or urgent care with influenza
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 313 | 98
Participants | 63 | 17

4. Secondary Outcome: Antibiotic Use
Description: Antibiotic use in children presenting to the ED or urgent care with influenza
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 313 | 98
Participants | 96 | 17

5. Secondary Outcome: Recurrent Visits
Description: Recurrent visits to the ED or healthcare provider in children presenting to the ED or urgent care with influenza
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 313 | 98
Participants | 21 | 4

6. Secondary Outcome: School Absenteeism
Description: Absenteeism from school or daycare in patients presenting to the ED or urgent care with influenza
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 313 | 98
Participants | 87 | 85

7. Secondary Outcome: Work Absenteeism
Description: Absenteeism from work in caregivers of children presenting to the ED or urgent care with influenza
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 313 | 98
Participants | 71 | 63

8. Other Pre Specified Outcome: Injectable Influenza Vaccine (IIV) Hospitalization
Description: Hospitalization among children who received IIV presenting to the ED or urgent care with influenza.
Time Frame: 0-14 days
Population: Outcome measure data is not required to be reported for this "other pre-specified" (not primary or secondary) outcome measure.
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days since enrollment until follow up
Description: Procedure related adverse events (nasal bleeding, nasal trauma from swab)
Arm/Group | Moderate-to-severe Influenza | Mild Influenza
All-Cause Mortality (participants affected / at risk) | 0/313 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/313 | 0/98
Other Adverse Events (participants affected / at risk) | 0/313 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02979626/Prot_SAP_000.pdf